CLINICAL TRIAL: NCT05955560
Title: Evaluating the Efficacy and Comfort of the PureWick Male External Catheter Against a Comparator in Healthy Volunteers
Brief Title: Male External Catheters' Comparison of Comfort and Efficacy
Acronym: MECCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UCC-23AC022
Record Dates: First submitted 2023-07-05; First posted 2023-07-21 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-06

CONDITIONS: Non-invasive Urine Output Management

STUDY DESIGN:
Intervention Model Description: Each subject acts as his own control, and therefore the difference in treatments is derived from a within-subject comparison.
Who Masked: Participant
Masking Description: Participants are blinded to which device is which and will remain blinded to treatment order until study completion. Investigator, Study Personnel and Sponsor will know which device the participant is treated with at any given time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Sequence 1 (Other): PureWick™ Male External Catheter is used first, followed by cross-over to Sage PrimoFit.
  Interventions: Device: PureWick Male External Catheter; Device: Sage PrimoFit
- Treatment Sequence 2 (Other): The Sage PrimoFit™ is used first, followed by cross-over to PureWick MEC.
  Interventions: Device: PureWick Male External Catheter; Device: Sage PrimoFit

INTERVENTIONS:
Device: PureWick Male External Catheter — The PureWick™ Male External Catheter (MEC) is intended for non-invasive urine output management in male patients. It is a single-use, non-sterile device. The PureWick™ Male External Catheter is a commercially available device which is Class I, 510(K) exempt.
  Other Names: PureWick MEC
Device: Sage PrimoFit — The PrimoFit External Urine Management for the Male Anatomy is indicated for the non-invasive external collection of urine for adult patients with male anatomy who require urine management. It is a single-use, non-sterile device. The Sage PrimoFit is a commercially available device which is Class I, 510(K) exempt.

SUMMARY:
A Prospective, Randomized, Crossover, Single-blind, Single Center Healthy Volunteer Study conducted over 1 day, with 2 voids using the PureWick (PW) Male external catheter (MEC) vs. comparator Sage PrimoFit™. This study is designed to assess the performance, comfort, and ease of use of the PW Male external catheter as compared to the comparator product.

DETAILED DESCRIPTION:
In this prospective, post-market, crossover, single-blind, single center healthy volunteer study, healthy males will be randomized 1:1 to a treatment sequence using two devices (PureWick™ Male External Catheter and Sage PrimoFit™) and followed for 1 day through 2 voids. Approximately 50 participants will be enrolled in this study to obtain 44 evaluable subjects. This study is designed to assess the performance, comfort, and ease of use of the PW Male external catheter.

The purpose of this study is to provide clinical evidence to compare the effectiveness and comfort of PureWick™ Male against a comparator for non-invasive urine output management in patients with varying male anatomy. Specifically, the study will collect data about how the male external catheters perform when participants are positioned on their side using a turning wedge with the head of the bed elevated, mimicking common patient positioning in the hospital setting.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Male Patient ≥ 18 years old
2. Male anatomy at time of enrollment
3. Ability to speak and understand English
4. Willing to comply with all study procedures in this protocol
5. Able to independently void urine
6. Provision of signed and dated informed consent form

Exclusion Criteria:

1. Urinary incontinence which does not allow the subject to spontaneously void
2. Frequent episodes of bowel incontinence
3. Has Urinary Retention
4. Has any irritation, wound, open lesion, at the application site, on the genitalia, perineum, or sacrum
5. Recent surgery of the external urogenital tract, penis, or pubic area
6. Not able to comply with study procedures independently without required assistance
7. Any other condition that, in the opinion of the investigator, would preclude them from participating in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Victoria Sena, RN, Principal Investigator — Tampa General Hospital
Locations (1):
- USF Health Center for Advanced Medical Learning and Simulation (CAMLS), Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were identified by a third party recruitment vendor. Targeted enrollment included 50 male, healthy volunteer participants in proximity to the clinical site. Participants were excluded if incontinent to urine or feces, or had any pre-existing wound, open lesion or irritation in the device application area.
Groups:
- PureWick Male, Then Sage PrimoFit: Participants used PureWick MEC for void 1. After consuming fluids to ensure adequate bladder volume, participants completed void 2 using Sage PrimoFit.
- Sage PrimoFit, Then PureWick Male: Participants used Sage PrimoFit for void 1. After consuming fluids to ensure adequate bladder volume, participants completed void 2 using PureWick MEC.
Period: Void 1
Arm/Group | PureWick Male, Then Sage PrimoFit | Sage PrimoFit, Then PureWick Male
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0
Period: Void 2
Arm/Group | PureWick Male, Then Sage PrimoFit | Sage PrimoFit, Then PureWick Male
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This single-blind, controlled, crossover study randomized participants 1:1 to a treatment sequence using two non-invasive urine collection devices (PureWick Male External Catheter or Sage PrimoFit). Participants were followed for 1 day through 2 voids. After void 1 was completed with PureWick MEC or Sage PrimoFit, participants consumed fluids and completed void 2 using the alternative device.
Arm/Group | All Study Participants
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of overall study population
  years | 40.8 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 30
  White | 22
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 59
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (8.58)

OUTCOME MEASURES:

1. Primary Outcome: Performance of the PureWick MEC Against an Established Comparator
Description: Capture rate following void (captured as % of urine captured by device and collected in canister, measured by weight).
  Prior to each void, the weight of the empty urine collection canister and the weight of a dry absorbent pad are collected. Participants void into the device while laying in a bed with the absorbent pad underneath them. After each void, the post-void weight of the urine collection canister and the post-void weight of the absorbent pad are collected.
  Capture rate is calculated as the weight of captured urine (post-void canister weight - pre-void canister weight) / total urine volume (captured urine (post-void canister weight - pre-void canister weight) + leaked urine (post-void pad weight - pre-void pad weight)) * 100.
Time Frame: Approximately 2 hours after device placement
Population: All enrolled and randomized participants were included in the primary endpoint efficacy analysis
Measure: Mean (Standard Deviation); unit: Percentage of urine captured
Arm/Group | PureWick Male External Catheter | Sage PrimoFit
Number analyzed (Participants) | 59 | 59
Percentage of urine captured
  Void 1: number analyzed (Participants) | 30 | 29
  Void 1 | 97.8 (10.03) | 90.7 (20.68)
  Void 2: number analyzed (Participants) | 29 | 30
  Void 2 | 91.1 (25.84) | 85.2 (21.67)
Statistical Analysis 1: Comparison: PureWick Male External Catheter vs Sage PrimoFit; Test type: Superiority; p = 0.04, t-test, 2 sided — A two-sided paired t-test was used and p-value derived. The threshold for statistical significance was p < 0.05

2. Secondary Outcome: Performance of the PureWick MEC in Morbidly Obese Subpopulation
Description: Capture rate following void (captured as % of urine captured by device and collected in canister, measured by weight).
Time Frame: Approximately 2 hours after device placement
Population: As there were only 2 participants that were assessed as unable to use traditional sheath style condom catheters, the secondary analysis was performed on the ITT subpopulation of morbidly obese participants.
Measure: Mean (Standard Deviation); unit: Percentage of urine captured
Arm/Group | PureWick Male External Catheter | Sage PrimoFit
Number analyzed (Participants) | 15 | 15
Percentage of urine captured
  Void 1: number analyzed (Participants) | 8 | 7
  Void 1 | 99.7 (0.88) | 83.5 (32.24)
  Void 2: number analyzed (Participants) | 7 | 8
  Void 2 | 80.8 (36.94) | 79.3 (23.32)

3. Secondary Outcome: Participant Comfort
Description: Overall comfort on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome, where 1 = Very Uncomfortable, 2 = Uncomfortable, 3 = Neither Comfortable or Uncomfortable, 4 = Comfortable, and 5 = Very Comfortable.
  The last survey question related to likelihood to recommend the device ranged from 1-5 with higher scores indicating a better outcome, where 1 = Very Unlikely, 2 = Unlikely, 3 = Neither Likely Nor Unlikely, 4 - Likely, and 5 = Very Likely.
Time Frame: Approximately 2 hours after device placement
Population: All enrolled and randomized participants were included in the secondary endpoint analysis (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick Male External Catheter | Sage PrimoFit
Number analyzed (Participants) | 59 | 59
score on a scale
  Device Placement Comfort | 3.85 (1.4) | 3.69 (1.34)
  Device Voiding Comfort | 3.71 (1.35) | 3.41 (1.23)
  Device Removal Comfort | 3.57 (1.11) | 3.62 (1.3)
  Likelihood to recommend device to a loved one | 3.98 (1.33) | 3.51 (1.5)

4. Secondary Outcome: Participant Comfort Scale Survey
Description: as for outcome 3
Time Frame: Approximately 2 hours after device placement
Population: ITT removing subjects who used source worksheet with typographic errors on Likert scale scoring choices
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick Male External Catheter | Sage PrimoFit
Number analyzed (Participants) | 38 | 38
score on a scale
  Device Placement Comfort | 4.29 (1.06) | 3.92 (1.24)
  Device Voiding Comfort | 4.0 (1.25) | 3.58 (1.27)
  Device Removal Comfort | 3.84 (1.0) | 3.92 (1.17)
  Likelihood to recommend device to a loved one | 3.97 (1.44) | 3.58 (1.54)

5. Secondary Outcome: Ease of Use by Health Care Professional (HCP)
Description: Ease of use score on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome, where 1 = Very Difficult, 2 = Somewhat Difficult, 3 = Average Difficulty, 4 = Somewhat Easy, and 5 = Very Easy.
Time Frame: Approximately 2 hours after device placement
Population: All enrolled and randomized participants were included in the secondary endpoint analysis (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick Male External Catheter | Sage PrimoFit
Number analyzed (Participants) | 59 | 59
score on a scale
  Ease of device placement | 4.59 (0.65) | 4.58 (0.7)
  Ease of device removal | 4.71 (0.56) | 4.81 (0.47)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | PureWick Male External Catheter | Sage PrimoFit
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

LIMITATIONS AND CAVEATS:
The secondary endpoint intended to assess capture rate in men with a buried penis/anatomy not compatible with a traditional sheath-style catheter; however, there were too few men meeting this criteria to make this assessment. Instead, the ITT subpopulation of morbidly obese participants was assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT05955560/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT05955560/SAP_001.pdf